CLINICAL TRIAL: NCT04238637
Title: Phase II Study of Immunotherapy With Durvalumab (MEDI4736) or Durvalumab and Tremelimumab, Both Combined With Y-90 SIRT Therapy in Advanced Stage Intrahepatic Biliary Tract Cancer (BTC)
Brief Title: Immunotherapy Combined With Y-90 SIRT Therapy in Advanced Stage Intrahepatic Biliary Tract Cancer (BTC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMUWHY
Record Dates: First submitted 2019-12-19; First posted 2020-01-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Bile Duct Cancer; Intrahepatic Biliary Tract Carcinoma; Intrahepatic Cholangiocarcinoma; BTC; iBTC; iCCA
MeSH Terms: conditions — Cholangiocarcinoma | interventions — durvalumab; tremelimumab; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Two randomized Treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Durvalumab
  Interventions: Drug: Durvalumab
- Arm 2 (Experimental): Durvalumab in combination with Tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous Infusion)
  Other Names: Other Name: MEDI4736
Drug: Tremelimumab — Tremelimumab IV (intravenous Infusion)
  Other Names: Study treatment
  Arms: Arm 2

SUMMARY:
A multicenter Phase II, randomized, prospective, open-label Trial investigating the clinical impact on combining Specific Internal Radiotherapy (SIRT) with the PD1-L Inhibitor Durvalumab and the CTLA-4 Inhibitor Tremelimumab in patients with intrahepatic Biliary Tract Cancer

DETAILED DESCRIPTION:
IMMUWHY Phase II Clinical Trial will test the Addition of the immunotherapeutic agents Durvalumab and Tremelimumab after an initial Standard of Care SIRT in patients suffering from non-resectable intrahepatic Biliary Tract Cancer. Patients will be randomized into two experimental arms, one receiving Durvalumab only, the other one receiving Durvalumab + Tremelimumab. Clinical Outcomes will be compared vs. historical datasets.

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent and locally required authorization (European Union [EU]: General Data Privacy Regulation (GDPR)) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years.
3. Histologically documented diagnosis of locally-advanced OR limited metasized intrahepatic BTC not amenable to curative treatment (tumor resection or ablation), specified as

   * Tumor being confined to the liver or
   * In case of presence of extrahepatic lesions, metastasis must be stable AND of limited extent* AND patient must have a potential benefit from study participation in comparison to standard of care systemic therapy per local tumor board evaluation.

     *Limited extent is defined in this protocol as presence of
     * EITHER ≤3 malignant extrahepatic lymph nodes (short axis diameter ≥3cm)
     * OR metastatic lesions in one organ other than liver (if only single lesion is present diameter MUST be < 3cm; if up to 3 lesions in one organ each lesion MUST be ≤ 1cm).
     * Presence of peritoneal or brain metastatsis excludes patients from study participation (see exclusion criterion #4)
   * Tumor tissue (block or at least 4 slides) is available for translational research.
4. Patients with prior chemotherapy and/or immunotherapy can be enrolled if ONE of the following criteria is met:

   * Capecitabin or gemcitabine+cisplatin in the adjuvant setting
   * Experienced progressive disease under gemcitabine+cisplatin therapy in the advanced setting
   * Stable disease after 3 months of gemcitabine+cisplatin treatment
   * Experienced progressive disease under durvalumab+ gemcitabine+cisplatin in first line treatment
   * Experienced progressive disease under pembrolizumab+ gemcitabine+cisplatin in first line treatment
5. Has been considered candidate for standard-of-care Y-90 SIRT therapy per Investigator decision and after prior consultation with the tumor board if available at site and does not display contraindications against SIRT.

   Contraindications against SIRT would be
   * hepatic tumor load > 50%
   * any Gastrointestinal deposition that cannot be corrected via angiographic techniques
   * irreversibly elevated serum bilirubin
   * renal insufficiency
   * increased pulmonary shunt fraction being able to deliver > 16.5 mCi to the lungs
   * gastrointestinal ulceration
   * hepatic dysfunction
   * biliary complications
   * portal hypertension
   * vascular injury and lymphopenia.
6. Performance status (PS) ≤ 1 (ECOG scale).
7. Body weight >30 kg
8. At least one measurable site of disease as defined by RECIST 1.1 criteria.
9. Adequate bone marrow and renal function
10. Adequate hepatic function (with stenting for any obstruction, if required)
11. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
13. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
14. Must have a life expectancy of at least 12 weeks.
15. If patient has concurrent Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection, meets the following criteria:

    * Patients with HBV or HCV infection should be monitored for viral levels during study participation.
    * Patients with detectable hepatitis B surface antigen (HBsAg) or detectable HBV DNA should have HBV DNA < 100 IU/ml and should be managed per local treatment guidelines.

Controlled (treated) hepatitis B subjects will be allowed if they started treatment at the time point of enrollment into the study by the latest and treatment is continued during study participation and for ≥ 6 months after end of study treatment.

- HCV patients with advanced BTC are mostly not treated for their HCV infection. However, patients treated for HCV are considered suitable for inclusion if antiviral therapy has been completed ≥ 30 days prior to first administration of study drug.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study.
2. Participation in another clinical study with an investigational product within 21 days prior to the first dose of the study treatment.
3. Prior immunotherapy or use of other investigational agents, including prior treatment with an anti-Programmed Death receptor-1 (PD-1), anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-cytotoxic T-lymphocyte associated antigen-4 (anti-CTLA-4) antibody, therapeutic cancer vaccines, apart from durvalumab and pembrolizumab as PD-L1 inhibitor in first line therapy.
4. Presence of peritoneal carcinomatosis or brain metastases.
5. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
6. Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (eg, hormone replacement therapy) is acceptable.
7. Prior radiotherapy treatment before the first dose of any study drug.
8. Major surgery (as defined by the Investigator) within 4 weeks prior to enrollment into the study; patients must have recovered from effects of any major surgery. Note: Local non-major surgery for palliative intent (e.g. surgery of isolated lesions, per-cutaneous biliary drainage or biliary stenting) is acceptable.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis].
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, , serious active, uncontrolled, gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
11. History of non-infectious pneumonitis requiring steroids, or patients with Grade ≥ 2 pneumonitis.
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
13. History of leptomeningeal carcinomatosis
14. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have a CT/ MRI of the brain prior to study entry.
15. History of active primary immunodeficiency
16. History of allogenic organ transplantation.
17. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), or human immunodeficiency virus (positive HIV 1/2 antibodies) or active hepatitis B/hepatitis C co-infection.
18. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab.
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of durvalumab.
20. Known allergy or hypersensitivity to any of the IMPs or any of the constituents of the product.
21. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
22. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
23. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].
24. Receipt of live attenuated vaccine within 30 days prior to the first administration of any of the IMPs and without need to receive any live attenuated vaccines during study conduct and for up to 30 days after end of Durvalumab treatment or 90 days after end of Tremelimumab treatment respectively.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate (ORR) according to RECIST 1.1 | 20 months
  Proportion of allocated subjects with best response of complete or partial response

SECONDARY OUTCOMES:
Safety (rate of adverse events) | From first patient included until study closure (approx. 43 months after First Patient Included)
  Type, incidence and severity of AEs and SAEs graded according to NCI CTCAE v5.0
Duration of response (DoR) | From first measurement of CR or PR per RECIST 1.1 until disease progression occurs (up to 43 months until Study Closure)
  Time from that the measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that the PD is objectively documented or death
Progression free survival (PFS) | From date of randomization until disease progression occurs (up to 43 months until Study Closure)
  Time from the date of randomization to the date of first observed disease progression (investigator assessment according to RECIST 1.1) or death from any cause
Overall Survival (OS) | Date of enrollment until date of death if applicable (up to 43 months until Study Closure)
  time from the date of treatment allocation to the date of death.

OTHER OUTCOMES:
Translational research | 3 months
  Exploratory: Predictive biomarkers that with a potential effect on Objective Response Rate, Duration of Response, Progression Free Survival and Overall Survival via blood sample collection + genetic subset analysis. The following translational research is currently planned, but may be adapted taking into account new research data: Tumors will be tested for mRNA expression of PD-1, PD-L1 and PD-L2 expression, Immune cell infiltrates (IGHM, CD3, CD8, FOXP3, CD68, CD205), Chemokines (CXCL9. CXCL10, CXCL13) and invasion markers (MMP7, MMP9)

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Professor, Study Director — IKF Klinische Krebsforschung GmbH
Locations (8):
- Germany (8):
  - University Hospital Dresden, Dresden
  - Clinic Essen Center, Essen
  - University Hospital Essen, Essen
  - University Hospital Halle, Halle
  - Hannover Medical School, Hanover
  - University Hospital Jena, Jena
  - Munich Clinic Bogenhausen, Munich
  - University Hospital Munich Grosshadern, Munich

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.